CLINICAL TRIAL: NCT00429078
Title: Phase I Trial of 2nd Generation Anti-CEA Designer T Cells in Gastric Cancer
Brief Title: Trial of 2nd Generation Anti-CEA Designer T Cells in Gastric Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3020-01A1
Record Dates: First submitted 2007-01-30; First posted 2007-01-31 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; T Cells; Gene Transfer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: 2nd Generation Designer T Cells

SUMMARY:
This study proposes to determine the safety and tolerability of 2nd generation designer T cells in patients with gastric cancer.Designer T cells are prepared by removing white blood cells from the participant, and then modifying these cells so that they recognize tumor antigen(CEA). These modified cells are then re infused back into the participant so that they can attack and kill tumor cells.Eligibility for this study is diagnosis of carcinoma of the stomach with failure to respond to standard curative therapy. Tumors must express CEA as demonstrated by elevated serum CEA >10ng/ml and be measurable radiologically or by physical exam.

DETAILED DESCRIPTION:
T cells can penetrate virtually every biologic space and have the power to dispose of normal or malignant cells as seen in viral and autoimmune diseases and in the rare spontaneous remissions of cancer. However, T cells are easily tolerized to self or tumor antigens and "immune surveil¬lance" has manifestly failed in every cancer that is clinically apparent. It is the goal of this study to supply the specificities and affinities to patient T cells without regard for their "endogenous" T cell receptor repertoire, directed by antibody-defined recognition to kill malignant cells based on their expression of antigen. We will achieve this by preparing chimeric IgCD28TCR genes in mammalian expression vectors to yield "designer T cells" from normal patient cells. Prior studies in model systems demonstrated that recombinant IgCD28TCR could direct modified T cells to respond to antigen targets with IL2 secretion, cellular proliferation, and cytotoxicity, the hallmarks of an effective, self-sustaining immune response. It therefore becomes of paramount interest to extend these studies to a human system of widespread clinical relevance to explore the clinical potential of this new technology. The target antigen for these studies is carcinoembryonic antigen (CEA), which is prominently expressed on tumors of the stomach, colon and rectum, breast, pancreas and other sites.

ELIGIBILITY:
Inclusion Criteria:

* CEA expressing Gastric Cancer/GE Junction (>10ng/ml)
* Must have measurable disease radiologically or by physical exam
* Must have failed potentially curative standard therapy
* Must be 18 years of age or older
* No serious concomitant disease

Exclusion Criteria:

* Prior investigational treatment
* Requiring systemic steroids
* Serious medical conditions
* Concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Junghans, PhD, MD, Principal Investigator — Roger Williams Hospital